CLINICAL TRIAL: NCT04684017
Title: Anlotinib Plus Etoposide and Carboplatin as First-line Treatment for Extensive-stage Small Cell Lung Cancer: A Single Arm Phase II Trial
Brief Title: Anlotinib Plus Etoposide and Carboplatin as First-line Treatment for Extensive-stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, Head of department, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KS2039
Record Dates: First submitted 2020-12-22; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2019-12

CONDITIONS: SCLC; Anlotinib
Keywords: SCLC; Anlotinib
MeSH Terms: interventions — anlotinib; Etoposide; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anlotinib plus etoposide and carboplatin (Experimental): Etoposide and carboplatin plus anlotinib for 4 cycles and anlotinib as maintenance therapy
  Interventions: Drug: Anlotinib hydrochloride; Drug: Etoposide; Drug: Carboplatin

INTERVENTIONS:
Drug: Anlotinib hydrochloride — anlotinib 10 mg/day orally (from days 1 to 14 in a 21-day cycle)
  Other Names: anlotinib
Drug: Etoposide — 100mg/m2 iv on days 1-3 every 21 days for 4 cycles
  Other Names: VP-16
Drug: Carboplatin — AUC 5 iv on day 1 every 21 days for 4 cycles

SUMMARY:
This is a phase II, open-label, single center study, aiming to investigate safety and efficacy of etoposide and carboplatin (administered intravenously) in combination with anlotinib (administered orally) in treatment-naive advanced NSCLC.

DETAILED DESCRIPTION:
Lung cancer can be divided into small cell lung cancer (SCLC) and non-small cell lung cancer (NSCLC), of which SCLC accounts for about 15%-20%.Because of the high degree of malignancy of SCLC, patients often lose the opportunity of surgical treatment due to metastasis at the time of admission. Traditional cytotoxic drugs can improve the prognosis of patients and life treatment, but the survival benefit is very limited.

Vascular targeted therapy is an important treatment strategy for metastatic lung cancer.Anlotinib hydrochloride is a multi-target receptor tyrosine kinase inhibitor that has significant inhibitory activity against angiogenesis related kinases such as VEGFR1/2/3, FGFR1/2/3, and other tumor related kinases such as PDGFR /, C-Kit, Ret, etc. (e.g., Met, FGFR1/2/3). An exploratory phase II study explored the efficacy of third-line single-drug therapy for ED-SCLC and found significant improvement in prognosis.

Based on the above status and research results, the purpose of this study was to explore the efficacy and safety of anlotinib hydrochloride combined with etoposide/carboplatin in first-line treatment of extensive small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. According to the 8th edition of the AJCC/UICC TNM staging system for NSCLC, patients with extensive stage SCLC confirmed by histology or cytology and are confirmed to have at least one measurable lesion according to RECIST 1.1.
2. Without active brain metastasis
3. Previously treated with ICIs with progressive disease.
4. Age ≥18 years and ≤75 years;
5. ECOG PS score: 0 to 1
6. The main organs function is normal, that is, the following criteria met: good hematopoietic function, defined as absolute neutrophil count ≥1.5×109 /L, platelet count≥100 ×109 /L, hemoglobin ≥90g/L [no blood transfusion or no erythropoietin (EPO) dependence within 7 days before enrollment]; biochemical test results should meet the following criteria: BIL < 1.25 times the upper limit of normal value (ULN); ALT and AST < 2.5 × ULN; in case of liver metastases, ALT and AST < 5 × ULN; Cr ≤1.5×ULN or creatinine clearance (CCr) ≥60ml/min; Coagulation function is good, INR and PT ≤1.5 times ULN; if the subject is receiving anticoagulant treatment, PT should be within the prescribed range of use of anticoagulant drugs;
7. Women of child-bearing age should agree to take contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study and within 6 months after the study; non-breast-feeding patients whose serum or urinary pregnancy test should be negative; male patients should agree to take contraceptive measures during the study and within 6 months after the study.
8. Patients are voluntarily enrolled into the study, sign the informed consent form and have good compliance.

Exclusion Criteria:

1. Subjects with active CNS metastases are excluded.
2. Non-small cell lung cancer.
3. With obvious hemorrhage symptom
4. Patients with many factors affecting oral medication, such as dysphagia, gastrointestinal resection, chronic diarrhea and intestinal obstruction.
5. Combined with other tumors at the time of initial diagnosis.
6. Patients who have previously participated in other clinical trials and have not yet terminated the trial.
7. Patients who have acute infection that difficult to control.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
PFS | Time from randomization to progression, assessed 9-11 months
  Time from enrollment to progression or death

SECONDARY OUTCOMES:
ORR | 6-9 weeks
  Patients who were assessed as partial response or complete response
OS | 13-15 months
  Time from enrollment to death of any cause
DCR | 6-9 weeks
  Patients who were assessed as partial response, complete response or stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang W, Deng P, Kong T, Zhang B, Qian F, Dong Y, Chen Y, Chen L, Liu D, Zhang Y, Yang H, Han B. Safety and efficacy of anlotinib in combination with standard chemotherapy as first-line treatment for extensive-stage small cell lung cancer: A multi-center, prospective study (ACTION-2). Lung Cancer. 2022 Nov;173:43-48. doi: 10.1016/j.lungcan.2022.09.003. Epub 2022 Sep 8. PMID 36116169